CLINICAL TRIAL: NCT01060787
Title: An Observational Bilateral Evaluation of Corneal Endothelial Cell Density in Subjects Who Have Had a Fluocinolone Acetonide Implant for at Least One Year
Brief Title: Evaluation of Corneal Endothelial Cell Density in Subjects Who Have Had a Fluocinolone Acetonide Implant
Status: Completed | Type: Observational
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 440
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Inflammation; Uveitis
MeSH Terms: conditions — Inflammation; Uveitis | interventions — Fluocinolone Acetonide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fluocinolone Acetonide 0.59 mg: Participants who have had the fluocinolone acetonide (FA) drug delivery system 0.59 mg surgically implanted in the ocular vitreous chamber of one (1) eye for at least one (1) year.
  Interventions: Procedure: Fluocinolone Acetonide 0.59 mg
- Fluocinolone Acetonide 2.1 mg: Participants who have had the fluocinolone acetonide (FA) drug delivery system 2.1 mg surgically implanted in the ocular vitreous chamber of one (1) eye for at least one (1) year.
  Interventions: Procedure: Fluocinolone Acetonide 2.1 mg

INTERVENTIONS:
Procedure: Fluocinolone Acetonide 0.59 mg — At a single visit bilateral endothelial microscopy will be performed to determine endothelial cell density.
  Other Names: Retisert
  Groups: Fluocinolone Acetonide 0.59 mg
Procedure: Fluocinolone Acetonide 2.1 mg — At a single visit bilateral endothelial microscopy will be performed to determine endothelial cell density.
  Other Names: Retisert
  Groups: Fluocinolone Acetonide 2.1 mg

SUMMARY:
Investigate the impact of the Fluocinolone Acetonide (FA) intravitreal implants

DETAILED DESCRIPTION:
Investigate the impact of the Fluocinolone Acetonide (FA) intravitreal implants on corneal endothelial cell density.

ELIGIBILITY:
Inclusion Criteria:

* Had the FA intravitreal implant (0.59 or 2.1 mg) in only one eye for at least one(1) year
* Able and willing to follow instructions
* Able and willing to provide informed consent

Exclusion criteria:

* Is monocular
* Has current or relevant medical history that would interfere with their participation in this study, based on the judgment of the Investigator
* Had bilateral FA intravitreal implants
* Has a history of any severe/serious ocular pathology or medical condition that could result in the subject's inability to complete the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects having the fluocinolone acetonide intravitreal implant (0.59 or 2.1 mg) in only one eye for at least one (1) year.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Corneal Endothelial Cell Density | 1 Visit
  Bilateral specular microscopy will be performed and endothelial cell density will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Valeant Pharmaceuticals/Bausch & Lomb
Locations (1):
- Ophthalmic Partners of Boston, Boston, Massachusetts, United States